CLINICAL TRIAL: NCT03254225
Title: Sixteen Weeks of Resistance Training in Hypertensive Elderly, Effects on Heart Rate Variability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Alessandra Medeiros, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP1844640
Record Dates: First submitted 2017-08-11; First posted 2017-08-18 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Hypertension
Keywords: Hypertension; Elderly; Resistance training; Heart rate variability
MeSH Terms: conditions — Hypertension | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance training (Experimental): Resistance training performed three times at week for 16 weeks, in 8 exercises for the main muscles, the protocol of 3 sets of 10 repetitions with intensity of 50% of 1 maximum repetition (MR).
  Interventions: Behavioral: Resistance training
- Control (No Intervention): in this arm, the group will remain sedentary for the same period of the experimental group, and they will be invited to engage on the raining program after the sedentary period

INTERVENTIONS:
Behavioral: Resistance training — Resistance training performed three times at week for 16 weeks, in 8 exercises for the main muscles, the protocol of 3 sets of 10 repetitions with intensity of 50% of 1 maximum repetition (MR).
  Arms: Resistance training

SUMMARY:
This study evaluates the inffluence of 16 weeks of resistance training on heart rate variability of hypertensive elderlies patients. All volunteers will be divided in two groups, one will participate in a protocol of sixteen weeks of resistance training, an the other will remain sedentary.

DETAILED DESCRIPTION:
This study evaluates the inffluence of 16 weeks of resistance training on heart rate variability using time and frequency-domains by ECG tracks. Will be assessed the blood pressure using the ambulatory blood pressure monitoring method of hypertensive elderly patients. All volunteers will be divided in two groups, one will participate in a protocol of sixteen weeks of resistance training prescribed with a relative workload of 50% of 1 maximal repetition, an the ontrol group will remain sedentary.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensives
* Age 60 to 80 years
* Nonactive

Exclusion Criteria:

* Orthopedic problems or other problem that prevented the exercises
* Change in drug treatment during protocol
* Absence in more than 25% of the exercise sessions

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Blood pressure change due to resistance training | 16 weeks
  Blood pressure will be measured by Ambulatorial Monitoring Blood Pressure before and after 16 weeks of intervention.

SECONDARY OUTCOMES:
Heart rate variability - Time domain - change due to resistance training | 16 weeks
  Heart rate variability will be collected by electrocardiogram before and after 16 weeks of intervention
Heart rate variability - Frequency domain - change due to resistance training | 16 weeks
  Heart rate variability will be collected by electrocardiogram before and after 16 weeks of intervention
Heart rate variability - Non-linear methods - change due to resistance training | 16 weeks
  Heart rate variability will be collected by electrocardiogram before and after 16 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Fabio T Montrezol, Principal Investigator — Federal University of São Paulo
Locations (1):
- Fabio Tanil Montrezol, Santos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No